CLINICAL TRIAL: NCT06043193
Title: Evaluation of the Quality of Life and Tolerance of Patients Treated With Vectorized Internal Radiotherapy (RIV) for a Neuro Endocrine Tumor (NET) in the Auvergne-Rhône-Alpes Region.
Acronym: AURA-RIV-TNE
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0367; 2023-A01344-41 (Other: ID-RCB)
Record Dates: First submitted 2023-08-10; First posted 2023-09-21 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Neuroendocrine Tumour
Keywords: IRV, Neuroendocrin, Quality of life
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Major subjects, suffering from metastatic neuroendocrine tumours: Major subjects, suffering from metastatic neuroendocrine tumours, for whom the indication for treatment by vectorized internal radiotherapy is decided in a multidisciplinary consultation meeting (National Reference Network for the management of Neuro-Endocrine Tumors) and who will be treated in one of the 5 centers in the AURA region

SUMMARY:
The study consists of having participants complete quality of life questionnaires (PROMs) at the time of the cures +/- one week and in the middle of the intercure time +/- one week.

As all the collection times do not correspond to a consultation or a visit to a medical service, The investigator wanted to develop a remote, computerized data collection solution.

Researchers have programmed an AURA-RIV-TNE care pathway (MOCAs: Engine for the organization and coordination of health acts) on the myHCL patient environment, taking up the course of the study presented in the form of a table in paragraph 6.2. Once the patient consents to participate in the study, he must create an account on the patient interface of his investigation center (myHCL, myCHUGA etc) as much as possible to facilitate data extraction.

Once the patient consents to participate in the study, the MOCAs AURA-RIV-TNE course will be associated with him in the Easily software, by defining the date week 0 (baseline) of the first treatment. This will allow automated sending of MAIL and SMS reminders at each questionnaire time. The MAILs will contain an internet link allowing the participant to be directly written to the questionnaires to be completed. A reminder system will be possible if the patient does not complete the questionnaire.

DETAILED DESCRIPTION:
The study consists of having participants complete quality of life questionnaires (PROMs) at the time of the cures +/- one week and in the middle of the intercure time +/- one week.

As all the collection times do not correspond to a consultation or a visit to a medical service, the investigator wanted to develop a remote, computerized data collection solution.

The investigator programmed an AURA-RIV-TNE care pathway (MOCAs: Engine for the organization and coordination of health acts) on the myHCL patient environment, taking up the course of the study presented in the form of a table in paragraph 6.2. Once the patient consents to participate in the study, he must create an account on the patient interface of his investigation center (myHCL, myCHUGA etc) as much as possible to facilitate data extraction.

Once the patient consents to participate in the study, the MOCAs AURA-RIV-TNE course will be associated with him in the Easily software, by defining the date week 0 (baseline) of the first treatment. This will allow automated sending of MAIL and SMS reminders at each questionnaire time. The MAILs will contain an internet link allowing the participant to be directly written to the questionnaires to be completed. A reminder system will be possible if the patient does not complete the questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Patient starting treatment with RIV validated in the RENATEN RCP;
* Patient having received written information about the study;
* Collection of the patient's non-objection
* Patients for whom treatment with RIV is administered within the framework of a clinical trial, may be included in the AURARIV-TNE study according to the written indications written in the 2 nd protocol of the sponsor of the clinical trial;
* Patients undergoing re-treatment with RIV can be included;

Exclusion Criteria:

* Persons deprived of their liberty by a judicial or administrative decision;
* Adults subject to a legal protection measure (guardianship, curatorship);

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subjects, suffering from metastatic neuroendocrine tumours, for whom the indication for treatment by vectorized internal radiotherapy is decided in a multidisciplinary consultation meeting (National Reference Network for the management of Neuro-Endocrine Tumors) and who will be treated in one of the 5 centers in the AURA region
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-03-20 (Actual); Study Completion 2026-09-20 (Estimated)

PRIMARY OUTCOMES:
The main quality of life criterion would be changed by the score of the EORTC-QLQC30 scale | Collection time: Week 0 (baseline) and 1 year
  The main quality of life criterion would be changed by the score of the EORTC-QLQC30 scale. 10% missing data tolerable

SECONDARY OUTCOMES:
Analysis of quality of life at baseline (week 0) | Collection time: Week 0 (baseline)
  Analysis of quality of life at baseline (Week 0) according to patient demographic profile and the characteristics of the tumour.
Analysis of the primary endpoint according to the Health Related Quality of Life (HRQoL) between inclusion, during the treatment and at 12 months. | Time of collection: Week 0 (baseline), 6 months and 1 year
  .Analysis of the primary endpoint according to the Health Related Quality of Life (HRQoL) between inclusion (before the first cycle-IVR1), during IVR (IVR2 to IVRn), at 6 and 12 months after IVR1, will be assessed by 4 questionnaires (EORTC QLQ-C30 + EORTC QLQ-GI.NET21 + EQ-5D + HADS) forming a composite criterion.and response to treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Saint-Etienne, Hôpital Nord, Saint-Priest-en-Jarez, Saint-Etienne
  - CH Métropole Savoie, Chambéry
  - Centre de Lutte Contre le Cancer Jean Perrin, Clermont-Ferrand
  - Hospices Civils de Lyon, Hopital Lyon Sud, Lyon

IPD SHARING:
Plan to Share IPD: No